CLINICAL TRIAL: NCT00597038
Title: A Phase I/II Study of Dasatinib and Dacarbazine in Patients With Metastatic Melanoma
Brief Title: A Phase I/II Study of Dasatinib and Dacarbazine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15256; 106128 (Other: USF IRB); CA180-092 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-05

CONDITIONS: Metastatic Melanoma
Keywords: Dasatinib; Dacarbazine
MeSH Terms: conditions — Melanoma | interventions — Dasatinib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I Dose Escalation (Experimental): Dasatinib and Dacarbazine (DTIC). The first cohort was a dasatinib dose of 50 mg by mouth (PO) twice a day (BID) given days 2-19 with DTIC given at a dose of 800 mg/m2 once every 3 weeks. The dose escalation was continued until MTD and a recommended Phase II dose was established.
  Interventions: Drug: Dasatinib and Dacarbazine (DTIC)
- Phase II Dose Treatment (Experimental): Dasatinib and Dacarbazine (DTIC). The recommended phase II dose was dasatinib 70 mg BID with dacarbazine 800 mgm^2.
  Interventions: Drug: Dasatinib and Dacarbazine (DTIC)

INTERVENTIONS:
Drug: Dasatinib and Dacarbazine (DTIC) — Arm A/ Phase I Potential Dose Levels.
  Dose Level -1: Dasatinib 40 mg; DTIC 600 mg/m^2. Dose Level 1: Dasatinib 50 mg; DTIC 800 mg/m^2. Dose Level 2: Dasatinib 70 mg; DTIC 800 mg/m^2. Dose Level 3: Dasatinib 70 mg; DTIC 1000 mg/m^2.
  Arm B/Phase II Potential Dose Levels.
  MTD1: Dasatinib 70 mg; DTIC 1000 mg/m^2. MTD2: Dasatinib 70 mg; DTIC 800 mg/m^2. MTD3: Dasatinib 100 mg: DTIC 1000 mg/m^2.
  Other Names: Sprycel (Dasatinib); DTIC (Dacarbazine)

SUMMARY:
The purpose of this study is to:

Phase I Objectives:

* Find the most tolerated dose to use for Phase II
* Collect information on how the body responds to this combination of study drug

Phase II Objectives:

* To determine the overall response of participants using this combination of study drug

The expression of proto-oncogene tyrosine-protein kinase (Src), a substance present in a significant proportion of melanomas plays a role in the growth, multiplying, and dividing of cancer cells. Melanoma cells appear to be sensitive to these agents that block the action of Src in concentrations that can be achieved in patients. We suggest that Src inhibitors (such as Dasatinib) may be a good choice for treatment of melanoma in combination with Dacarbazine (a chemotherapy drug that can cause the shrinkage of melanomas). We wish to to evaluate the Src inhibitor Dasatinib in combination with the chemotherapy drug Dacarbazine. The novel oral Src inhibitor Dasatinib may be able to increase the effectiveness of chemotherapy for melanoma compared to chemotherapy alone. Dacarbazine is a standard treatment for melanoma currently. The effectiveness of this chemotherapy drug may be increased by combination with Dasatinib. Dacarbazine has been approved by the US Food and Drug Administration (FDA) for treating melanoma; Dasatinib has been approved by the FDA to treat leukemia, but it has not been approved alone or in combination with Dacarbazine to treat melanoma.

DETAILED DESCRIPTION:
Patient will receive Dacarbazine intravenously (IV), which means it is given through a needle in a vein in the arm or through a venous port (if patient already has one). Dasatinib will be given orally starting day 2 for 17 days straight (days 2 through 19) starting the day after patient receives their first dose of Dacarbazine. The therapy will be repeated every 21 days (21 days = 1 cycle). Patient may be given other drugs before each cycle to help reduce side effects of the therapy. If patient experiences severe side effects, the amount of Dacarbazine and/or Dasatinib they receive in future cycles may be decreased.

Cycle 1 day 1:

* Dacarbazine Intravenous
* Toxicity assessment - evaluation of any side effects that patient may be experiencing
* Medical history*
* Physical examination* - measure height, weight, blood pressure, pulse, breathing rate, temperature, assessment of patient's energy and activity level (Eastern Cooperative Group [ECOG] Performance Status)
* Blood tests (3 tablespoons) for safety tests*- Complete blood count with differential and platelets (CBC), Comprehensive metabolic profile (CMP), & Magnesium test *(certain tests may not need to be performed if they were performed during screening within 1 week; study doctor will tell patient if they need to have these tests redone)

Cycle 1 day 8:

* Toxicity assessment - (these will be done for the first cycle of treatment, but will be discontinued for later cycles unless deemed necessary by study doctor)
* CBC - (1 tablespoon) (this will be done for the first cycle of treatment, but will be discontinued for later cycles unless deemed necessary by study doctor)
* Dasatinib orally

Cycle 1 day 15:

* Toxicity assessment - (these will be done for the first cycle of treatment, but will be discontinued for later cycles unless deemed necessary by study doctor)
* CBC - (1 tablespoon) these will be done for the first cycle of treatment, but will be discontinued for later cycles unless deemed necessary by study doctor)
* Dasatinib orally
* Blood sample for pharmacokinetic (PK) analysis

Patient will also take Dasatinib orally as instructed days: 2, 3, 4, 5, 6, 7, 9, 10, 11, 12, 13, 14, 16, 17, 18, 19 each cycle.

Day 1 for all cycles after the first cycle:

* Dacarbazine Intravenous (IV)
* Dasatinib orally
* Medical history
* Physical examination: measure height, weight, blood pressure, pulse, breathing rate, temperature, assessment of patient's energy and activity level (ECOG Performance Status)
* Blood tests (2 tablespoon) for safety tests: CMP & CBC
* An electrocardiogram (EKG)
* Computed tomography (CT) scan (done every other cycle starting with cycle 2)
* Toxicity assessment

If patient decides not to continue participation in this study or is taken off the study by their study doctor or the sponsor they will return to the clinic for one more visit.

During this visit the following procedures will be performed:

* Medical history
* Perform a physical examination: measure height, weight, blood pressure, pulse, breathing rate, temperature, assessment of patient's energy and activity level (Eastern Cooperative Group [ECOG] Performance Status)
* Blood tests (2 tablespoons) for safety tests: CBC & CMP
* Toxicity assessment Patient will need to take their assigned Dasatinib dose twice daily. It may be taken with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven melanoma with Stage IV or unresectable stage III disease
* Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 grade ≤1.
* Adequate organ function as defined by the following criteria:

  * Serum aspartate transaminase (AST); serum glutamic oxaloacetic transaminase (SGOT) and serum alanine transaminase (ALT); serum glutamic pyruvic transaminase (SGPT) ≤2.5 x local laboratory upper limit of normal (ULN), or AST and ALT less than or equal to 5 x ULN if liver function abnormalities are due to underlying malignancy
  * Total serum bilirubin ≤1.5 x ULN
  * Absolute neutrophil count (ANC) ≥1500/µL
  * Platelets ≥100,000/µL
  * Hemoglobin ≥9.0 g/dL (may be transfused or erythropoietin treated)
  * Serum calcium ≤12.0 mg/dL
  * Serum creatinine ≤1.5 x ULN
* Patients with CNS metastasis must have had either; a) resected central nervous system (CNS) metastasis without evidence of recurrence for >12 weeks; b) Brain metastasis treated by stereotactic radiosurgery without evidence of recurrence or progression for 12 weeks; Or, c) Multiple brain lesions treated with whole-brain radiation therapy (WBRT) with stable disease off corticosteroids for at least 12 weeks prior to start of therapy; and, d)Without any evidence of leptomeningeal disease. Patients must be neurologically intact.
* May have previous adjuvant therapy with interferon, vaccines or therapy with IL-2 or GM-CSF
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria is required in the Phase II portion of the trial. In the phase I part of the trial patients with evaluable but not measurable disease may be allowed with the permission of the Principal Investigator (PI)
* Eastern Cooperative Oncology Group (ECOG) PS 0-2

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks of starting the study treatment.
* NCI CTCAE grade 2 or greater hemorrhage within 4 weeks of starting the study treatment.
* History of or known carcinomatous meningitis, or evidence of symptomatic leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2.
* QTc >470 msec on baseline EKG.
* Hypertension that cannot be controlled by medications (>150/100 mm Hg despite optimal medical therapy).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or other active infection
* Ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg orally (po) daily for thromboembolism prophylaxis is allowed).
* Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* May not have had previous treatment with a Dacarbazine (DTIC) or temozolomide based chemotherapy regimen. In the Phase II part of the trial patients may not have had treatment with any chemotherapy regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, M.D.. Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Adil Daud, M.D., Study Chair — Helen Diller Family Comprehensive Cancer Center, University of California, San Francisco
Locations (2):
- United States (2):
  - Helen Diller Family Comprehensive Cancer Center, University of California, San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients had unresectable stage III or stage IV melanoma. Patients were required to have measurable or evaluable disease and prior treatment with dacarbazine or temozolomide was not allowed.
Groups:
- Phase I Dose Escalation: Dasatinib and Dacarbazine (DTIC). Dasatinib and Dacarbazine (DTIC). The first cohort was a dasatinib dose of 50 mg by mouth (PO) twice a day (BID) given days 2-19 with DTIC given at a dose of 800 mg/m2 once every 3 weeks. The dose escalation was continued until MTD and a recommended Phase II dose was established.
- Phase II Dose Treatment: Dasatinib and Dacarbazine (DTIC). Dasatinib and Dacarbazine (DTIC). The recommended phase II dose was dasatinib 70 mg BID with dacarbazine 800 mgm^2.
Period: Overall Study
Arm/Group | Phase I Dose Escalation | Phase II Dose Treatment
Started | 16 | 34
Completed | 14 (One did not complete due to PI decision, one did not complete due to progressive disease.) | 30 (Two patients withdrew, one did not complete due to progressive disease, one patient died.)
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation | Phase II Dose Treatment | Total
Number analyzed (Participants) | 16 | 34 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 20 | 26
  >=65 years | 10 | 14 | 24
Age, Continuous [Mean (Full Range); unit: years] | 68.1 [47 to 81] | 60.3 [34 to 80] | 62.3 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 10 | 21 | 31
Region of Enrollment [Number; unit: participants]
  United States | 16 | 34 | 50

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose
Description: To determine the maximum tolerated dose of dasatinib twice a day when given with dacarbazine. Adverse events were graded using Common Terminology Criteria for Adverse Events version 3.0. Dose-limiting toxicities are defined as any grade 4 haematological toxicity (except asymptomatic grade 4 neutropenia for =/< 7 days); prolonged grade 3 or 4 thrombocytopenia (47 days) or thrombocytopenia associated with bleeding, requiring platelet transfusion; any grade 3 or 4 nonhaematological toxicity despite optimal supportive care; any toxicity considered unacceptable by the study principal investigator.
Time Frame: 1 Year 3 Months
Population: All participants in Arm A
Measure: Number; unit: mg
Groups:
- Phase I Dose Escalation: Dasatinib and Dacarbazine (DTIC)
Arm/Group | Phase I Dose Escalation
Number analyzed (Participants) | 16
mg
  Recommended Dasatinib Dose mg | 70
  Recommended Dacarbazine Dose mg/m^2 | 800

2. Primary Outcome: Phase II - Number of Participants With Overall Response (OR)
Description: Phase II - To determine the overall response rate (ORR) of the combination of dasatinib and DTIC by the Response Evaluation Criteria in Solid Tumors (RECIST v1.0). Tumor assessments were made at baseline and at the end of every second cycle (i.e. every 6 weeks). Partial and complete responses were defined by the best treatment response achieved.
Time Frame: 1 Year 6 Months
Population: Patients receiving dasatinib at 70 mg PO BID
Measure: Number; unit: participants
Groups:
- Phase II Dose Treatment: Dasatinib and Dacarbazine (DTIC)
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 29
participants | 4

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) at 6 Months
Description: Phase II - PFS Rate in patients receiving dasatinib 70 mg orally (PO) twice a day (BID). Tumor assessments were made at baseline and at the end of every second cycle (i.e. every 6 weeks). Partial and complete responses were defined by the best treatment response achieved. Stable disease was defined as maintenance of the sum of lesions diameters between a 30% reduction and a 20% increase of overall tumour size over 12 weeks or longer.
Time Frame: 6 Months
Population: Patients receiving dasatinib at 70 mg PO BID
Measure: Number; unit: participants
Arm/Group | Phase II Dose Treatment
Number analyzed (Participants) | 29
participants | 6

4. Secondary Outcome: Number of Participants With 12 Month Overall Survival (OS)
Description: Phase II - To determine Overall Survival of patients treated with the combination of dasatinib and DTIC at 12 months.
Time Frame: 12 Months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Phase I Dose Escalation | Phase II Dose Treatment
Number analyzed (Participants) | 16 | 34
participants | 9 | 8

ADVERSE EVENTS:
Time Frame: First on treatment date to last off study date: 2 years, 4 months.
Arm/Group | Phase I Dose Escalation | Phase II Dose Treatment
Serious Adverse Events (participants affected / at risk) | 9/16 | 11/34
Other Adverse Events (participants affected / at risk) | 4/16 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation (N=16) | Phase II Dose Treatment (N=34)
Blood/Bone Marrow - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin - Grade 4 (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Neutrophils/granulocytes - Grade 4 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelets - Grade 3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelets - Grade 4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac general - Grade 3 (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 0 (0) | 1 (1)
Death not associated with CTCAE term - Disease progression not otherwise specified (NOS) - Grade 5 (General disorders) | 1 (1) | 2 (2)
Diarrhea - Grade 3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI - Lower GI NOS - Grade 3 (General disorders) | 0 (0) | 1 (1)
Hemorrhage, GI - Lower GI NOS - Grade 4 (General disorders) | 1 (1) | 0 (0)
Febrile neutropenia - Grade 3 (Infections and infestations) | 2 (2) | 1 (1)
Infection with Grade 3 or 4 neutrophils - skin - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - skin - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC - Joint - Grade 3 (Infections and infestations) | 1 (1) | 0 (0)
Edema - limb - Grade 3 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mental status - Grade 4 (Psychiatric disorders) | 0 (0) | 1 (1)
Pain - Abdomen NOS - Grade 3 (General disorders) | 0 (0) | 1 (1)
Pain - Abdomen NOS - Grade 4 (General disorders) | 1 (1) | 0 (0)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dyspnea - Grade 5 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Escalation (N=16) | Phase II Dose Treatment (N=34)
Allergic reaction/hypersensitivity - Grade 2 (General disorders) | 1 (1) | 0 (0)
Hemoglobin - Grade 2 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ascites (non-malignant) - Grade 2 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea - Grade 2 (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infection - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin - Grade 2 (Infections and infestations) | 1 (1) | 0 (0)
Pain - Chest wall - Grade 2 (General disorders) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No